CLINICAL TRIAL: NCT03408509
Title: Cognitive Training to Promote Brain Health: Implementation and Engagement
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: University of Dublin, Trinity College (Other); Global Brain Health Institute (GBHI) (Other)
Responsible Party: Principal Investigator, Rogerio Panizzutti, Associate Professor, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GBHI_ALZ-18-544160
Record Dates: First submitted 2018-01-12; First posted 2018-01-24 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Aging; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive training (Experimental)
  Interventions: Behavioral: Computerized cognitive training

INTERVENTIONS:
Behavioral: Computerized cognitive training — Posit Science Inc. will supply the software for the computerized cognitive training through the platform BrainHQ, which is available on line. The training program consists of a set of computerized exercises designed to improve the speed and accuracy of sensory information processing while engaging neuromodulatory systems involved in attention and reward. The rationale is that, in order to understand and remember information, the brain must first generate precise and reliable neurological responses that represent the sensory stimuli. These exercises continuously adjust the difficulty level to user performance to maintain an approximately 85% rate of correct responses. Trials with correct responses are rewarded with points and animations. The goal is to increase the effectiveness with which these stimuli engage and drive plastic changes in brain systems. Engagement is monitored by electronic data upload following each training session.

SUMMARY:
Cognition encompasses memory, attention, language and other brain capacities that are necessary for good quality of life and independence. Age-related cognitive decline starts at the third decade of life and in some cases can start to impact daily functioning in the late forties. Dementia is the most devastating consequence associated with age-related cognitive decline. Recent studies indicate that improving cognition by means of intensive computerized brain training can mitigate some aspects of agerelated cognitive decline, and may even have a role in preventing or delaying dementia onset. Critically, the capacity of a given individual to improve their cognitive performance after training is fundamentally related to engagement with the exercises. Currently, little is known about how to apply intensive computerized cognitive training effectively in the health system, ensuring engagement and best progress. This project aims to tackle this challenge by developing, applying and testing personalized approaches to implement cognitive training in daily life of older adults that were recently evaluated at Memory Clinics and their care partners. The community readiness approach will be implemented using semi-structured interviews, conducted with subjects that may be interested in cognitive training, key informant, and key stakeholders. Using this information, the investigators will design an individualized training program and follow up its application in a feasibility trial. Twenty participants, recently evaluated at different Memory Clinics in Ireland, will be recruited, interviewed and invited to engage, over the ensuing 2 to 3 months, in computerized cognitive training. Subjects will be assessed after completion of the intervention for training adherence and individual gains on the computerized exercises. In order to gain insight about regional specificities of the approach the investigators will perform a parallel project using the same methodology in Brazil. This project is expected to inform the future implementation of cognitive training in public health policies for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Being evaluated at a memory clinic in the last year, or be the care partner of a person evaluated at a memory clinic
* Adequate visual and auditory acuity to allow practice on the computerized training exercises
* Physical ability sufficient to allow performance of the computerized training exercises
* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Any medical condition that precludes performing the computerized training exercises
* Advanced dementia.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Engagement | 3 months
  will be defined as a continuous variable (number of hours of training completed by the participant).

SECONDARY OUTCOMES:
Individual gains on the computerized exercises | 3 months
  The computerized cognitive training platform, called BrainHQ, provided by Posit Science Inc, provides one measure of the individual gains on the computerized exercises with training.
Quantitative measure of motivation with the computerized training exercise | 3 months
  Motivation will be assessed by the quantitative score provided by the Adapted Ultrech Engagement Scale - UWES. The Utrecht Engagement Scale has 17 items that are scored on a 7-point Likert scale indicating the frequency with which engagement at a given activity happens in the situations described in each item (0 indicates "never" and 6 "always"). The factors Vigor and Concentration have six items each and the factor Dedication has 5 items. The final score of the Engagement corresponds to the sum of the scores on the three factors.
Qualitative motivation with the computerized training exercise | 3 months
  Qualitative motivation will be assessed using semi-structured interview.
Training adherence (dichotomic variable) | 3 months
  Training adherence will be defined as training more than 10 hours

CONTACTS AND LOCATIONS:
Locations (1):
- St James Hospital, Dublin, Ireland